CLINICAL TRIAL: NCT05127837
Title: Development of an Artificial Intelligence- Informed Digital Tool to Help Clinicians Practice Cognitive Behavioral Therapy for Psychosis (CBTp)
Brief Title: CBTpro: Scaling up CBT for Psychosis Using Simulated Patients and Spoken Language Technologies
Acronym: CBTpro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Lyssn.io, Inc. (Industry)
Responsible Party: Principal Investigator, Sarah Kopelovich, Associate Professor of Psychiatry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00014706; 5R42MH123215-02 (NIH)
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Psychosis; Schizophrenia; Schizo Affective Disorder; Bipolar Disorder; Depressive Disorder
Keywords: Clinician Training; AI (artificial Intelligence); Machine learning; NLP (natural language processing); Cognitive Behavioral Therapy (CBT)
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Bipolar Disorder; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as Usual (TAU) (No Intervention): CBT for psychosis distance learning course.
- CBTpro (Experimental): In addition to TAU, clinicians and clients receive the CBTpro training.
  Interventions: Behavioral: CBTpro

INTERVENTIONS:
Behavioral: CBTpro — CBTpro is a novel spoken language technology tool to support high-quality skills training in CBT for psychosis.
  Arms: CBTpro

SUMMARY:
The primary objective of this grant is to develop and evaluate an Artificial Intelligence-based clinical training tool--CBTpro--to support high-quality skills training in CBT for psychosis (CBTp). CBTpro will provide a rapid means of scaling and sustaining high-quality CBTp in routine care settings across the US.

DETAILED DESCRIPTION:
This fast-track Small Business Technology Transfer (STTR) grant is a partnership between the University of Washington and private company LYSSN that includes the development and iterative testing of CBTpro, a Computerized Clinician Support Tool designed to teach behavioral health providers and students Cognitive Behavioral Therapy for psychosis (CBTp). CBTpro uses natural language processing to provide automated speech-to-text and machine learning to score trainee's responses to simulated patients with psychosis.

Once technical reliability of the tool is achieved through iterative modifications based on usability and field trials, a randomized control trial will be conducted to assess CBTpro training vs. training as usual with N=100 providers / N=300 clients on clinician skills and client outcomes.

ELIGIBILITY:
Client Inclusion: Adults who speak English, meet with their provider who is participating in the study at least bi-weekly (2x a month), and do not plan to leave services in the next 6 months. Qualifying diagnoses for clients include: schizophrenia; schizoaffective disorder; schizophreniform disorder; delusional disorder; other specified schizophrenia spectrum and other psychotic disorder; unspecified schizophrenia spectrum or other psychotic disorder; bipolar disorder with psychotic features; major depressive disorder with psychotic features

Exclusion criteria: Dx of psychosis secondary to substance intoxication

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Change in Green Paranoid Thoughts Scale (GPTS) Total Score | 0,3,6 months
  The Green Paranoid Thoughts Scale (GPTS) is a 32-item self-report questionnaire designed to assess paranoid ideation over the past month. It consists of two 16-item subscales: Part A: Ideas of Social Reference and Part B: Persecutory Ideas. Each item is rated on a 5-point Likert scale from 1 ("Not at all") to 5 ("Totally"). Subscale scores range from 16 to 80, and the total score ranges from 32 to 160, with higher scores indicating more severe paranoid thinking. A reduction in total or subscale scores indicates improvement in paranoid ideation.

SECONDARY OUTCOMES:
Change in CHOICE-SF (Choice of Outcome in CBT for Psychosis- Short Form) | 0,3,6 months
  The CHOICE-SF is a 12-item self-report questionnaire designed to assess perceived progress toward recovery among individuals receiving cognitive behavioral therapy for psychosis (CBTp). Each item is rated on a scale from 0 ("Not at all") to 10 ("Extremely") with the exception of the final question which is open-entry. Total scores range from 0 to 110, with higher scores reflecting greater perceived progress in psychological recovery. An increase in the CHOICE-SF score indicates improvement in recovery; a decrease suggests reduced perceived progress.
Change in in Sheehan Disability Scale (SDS) Total Score | 0,3,6 months
  The Sheehan Disability Scale (SDS) is a 3-item self-report measure that assesses functional impairment in three domains: work/school, social life, and family life/home responsibilities. Each item is rated on an 11-point scale from 0 ("Not at all impaired") to 10 ("Extremely impaired"). The total score ranges from 0 to 30, with higher scores indicating greater functional impairment. A decrease in the total score reflects improved functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kopelovich, PhD, Principal Investigator — University of Washington
Locations (13):
- United States (13):
  - South Central Health and Rehabilitation Programs, Los Angeles, California
  - Psynergy, Morgan Hill, California
  - Telecare, San Jose, California
  - Integrated Services of Kalamazoo, Kalamazoo, Michigan
  - Community Mental Health Authority of Clinton, Eaton, and Ingham Counties (CEICMH), Lansing, Michigan
  - Coleman Health Services, Akron, Ohio
  - PeaceHealth, Eugene, Oregon
  - Cascadia, Portland, Oregon
  - Lifeworks NW, Portland, Oregon
  - Harborview Medical Center, Seattle, Washington
  - Sound Health, Seattle, Washington
  - Frontier Behavioral Health, Spokane, Washington
  - Comprehensive Healthcare, Yakima, Washington

IPD SHARING:
Plan to Share IPD: Yes
Research subject's de-identified data will be shared through the National Institute of Mental Health Data Archive (NDA).